CLINICAL TRIAL: NCT00532350
Title: A Randomized, Double-blind, Placebo-controlled Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of an Efficacious Dose of QAT370 Compared to Open-label Tiotropium Bromide Following Once Daily Dosing for 7 Days in COPD Patients
Brief Title: Safety and Tolerability QAT370 Compared to Tiotropium in Patients With Chronic Obstructive Pulmonary Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: External Affairs, Novartis
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CQAT370A2103
Record Dates: First submitted 2007-09-19; First posted 2007-09-20 (Estimated); Last update posted 2020-12-19 (Actual); Status verified 2010-09

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; pharmacokinetics; plethysmography; cycle ergometry; exercise testing; spirometry
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Tiotropium Bromide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): QAT370
  Interventions: Drug: QAT370
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- 3 (Active Comparator): Tiotropium
  Interventions: Drug: Tiotropium

INTERVENTIONS:
Drug: QAT370
  Arms: 1
Drug: Placebo
  Arms: 2
Drug: Tiotropium
  Arms: 3

SUMMARY:
This study will assess the safety and tolerability of QAT370 compared to tiotropium in patients with COPD.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 40 and 80 years of age with controlled COPD.
* Women must be surgically sterilized or postmenopausal. Additional birth control and post-menopausal information will be available at time of enrollment.
* Body mass index (BMI) must be within the range of 18 to 32 kg/m2

Exclusion Criteria:

* Participation in any interventional clinical investigation with 4 weeks of study start
* Blood loss or donation of 400 mL or more within 2 months of study start Significant illness (other than respiratory) within 2 weeks of study start
* Past medical personal or close family history of clinically significant ECG abnormalities
* Any medical condition that may interfere with exercise testing or that may make spirometry unsafe
* A known hypersensitivity to the drug.
* History of immunocompromise, including a positive HIV test result.
* History of drug or alcohol abuse within 12 months of study start
* Any condition that may compromise patient safety

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2007-07; Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Forced expiratory volume in 1 second | Days 1 and 7

SECONDARY OUTCOMES:
Forced expiratory volume in 1 second and corresponding parameters for inspiratory capacity. | Days 1 and 7

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Principal Investigator — Investigative site
Locations (3):
- Germany (3):
  - Novartis investigative site, Berlin
  - Novartis Investigative site, Mannheim
  - Novartis Investigative site, Wiesbaden

REFERENCES:
- See also: Results for CQAT370A2103 can be found on the Novartis Clinical Trial Results Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=2637